CLINICAL TRIAL: NCT02832271
Title: Randomised Double-blinded Placebo Controlled Trial of Green Tea Extract for Endometriosis
Brief Title: Green Tea Extract for Endometriosis Treatment
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other); Sun Yat-sen University (Other); Guangdong Provincial Hospital of Traditional Chinese Medicine (Other); Jiangxi University of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, Ronald Wang, Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 6904267
Record Dates: First submitted 2016-07-05; First posted 2016-07-14 (Estimated); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Endometriosis
MeSH Terms: conditions — Endometriosis | interventions — Tea

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- green tea group (Active Comparator): green tea extract SUNPHENON EGCg for women with ultrasound confirmed endometriosis
  Interventions: Drug: SUNPHENON EGCg
- placebo group (Placebo Comparator): placebo fro women with ultrasound confirmed endometriosis
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SUNPHENON EGCg — SUNPHENON EGCg Oral, 400mg, twice per day
  Other Names: green tea extract
  Arms: green tea group
Drug: Placebo — Placebo
  Arms: placebo group

SUMMARY:
The purpose of the study is to evaluate the efficacy and safety of green tea in endometriosis.

DETAILED DESCRIPTION:
Women with endometrioma will be randomised into either the experimental group or the placebo comparator group in a 1:1 ratio. The subjects will be given SUNPHENON EGCg or placebo for 3 months prior to their planned surgery.

ELIGIBILITY:
Inclusion Criteria:

* Complaints of pelvic pain, dysmenorrhoea and/or dyspareunia ≥ 6 months; and
* Verbal pain rating scale > 4/10 and visual analogue pain scale > 4cm; and
* Ultrasound confirmed endometrioma with or without fibroid and adenomyoma; and
* Planned surgery treatment within 4-6 months

Exclusion Criteria:

* Age < 20 years beyond or >40 year behind the active reproductive age; or
* BMI <18.5 kg/m2 as underweight or >25 kg/m2 as overweight; or
* Chronic pelvic pain or low back pain due to other medical conditions, e.g. urological disorders and orthopaedic disorders; or
* Secondary dysmenorrhoea due to gynaecological conditions other than endometriosis, e.g. pelvic inflammatory diseases, genitourinary infections, gynaecological tumours, etc.; or
* Primary dysmenorrhoea without any underlying disease identified; or
* Ultrasound suggested polycystic ovary, haemorrhagic ovarian cyst, ovarian dermoid cyst, cystic neoplasm, tubo-ovarian abscess or other ovarian pathologies in the same ovary; or
* Chronic medical conditions under long-term medications; or
* Endometriosis under active medication in past 1 month; or
* History of herbal medicine intake in past 1 month

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 185 (Actual)
Dates: Start 2016-12-08 (Actual); Primary Completion 2022-12 (Actual); Study Completion 2022-12 (Actual)

PRIMARY OUTCOMES:
Change in endometriotic lesion size | At 0 and 3 months of treatment
  Structural MRI will be performed with a 3T whole-body clinical scanner by a radiologist. The total volume of endometriotic mass in the endometrioma indicated by the positive enhanced image will be quantified. The endometriotic mass before treatment will be used as baseline for comparison and analysis. Prior to the planned surgery, another structural MRI will be performed again to assess the changes in endometriotic mass after treatment.

SECONDARY OUTCOMES:
Changes in pain scores assessed by ESS and VAS | At 0, 1.5 and 3 months of treatment
  The severity of the pain will be quantified and evaluated by an Endometriosis Symptom Severity verbal rating scale (ESS). With ESS, subjects will rate their pain from score 0 as absence of pain to 10 as the most severe intolerable pain. A modified Biberoglu-Behrman 10cm visual analogue scale (VAS) will also be used to evaluate the pain experienced by the subjects. For VAS, subjects will mark the level of pain that they encounter on a graphic scale which range from 0cm as absence of pain to 10cm as the pain becomes as bad as it could possibly be. The 2 measurements will be recorded separately.
Changes in quality of life assessed by SF36 | At 0, 1.5 and 3 months of treatment
  Quality of life will be assessed using the standard SF36 instrument. SF36 consists of a medical survey which consists of 8 domains. The domain scores are rated onto a scale from 0 as worst health to 100 as best health. The Endometriosis Health Profile version 5 (EHP5) will as well be used to assess the quality of life. EHP5 contains 5 core and 6 modular questionnaires. Each item is rated on a 5-point scale (from 0=never to 4=always). The overall score will be transformed to a scale of 0 as best health and 100 as worst health.
Change in endometriotic growth assessed by pathology | At 0 and 3 months of treatment
  Endometriotic cysts biopsies will be collected during the surgery. Endometriotic growth will be confirmed by the presence of endometrial epithelial glands and stroma in the biopsies. The biopsies will be compared to the endometriotic mass before treatment.
Change in total number of neovasculatures assessed by DCE-MRI | At 0 and 3 months of treatment
  Subjects will undergo pelvic DCE-MRI for measurement of the total number of neovasculatures in the endometriotic mass.
Change in density of neovasculatures assessed by DCE-MRI | At 0 and 3 months of treatments
  Subjects will undergo pelvic DCE-MRI for measurement of the density of neovasculatures in the endometriotic mass.
Number of Participants with adverse outcome and side effects | At 0, 1.5 and 3 months of treatment
  any related and unrelated severe adverse events and adverse events, side-effects

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Wang, MD PhD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Shatin, Hong Kong

IPD SHARING:
Plan to Share IPD: No